CLINICAL TRIAL: NCT03972189
Title: Phase II, Open Label, Single Arm Study of the Efficacy and Safety of TQ-B3101 in Patients With ROS1-positive Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Safety and Efficacy Study of TQ-B3101 in Patients With ROS1-positive Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3101-II-01
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: ROS1-positive Non-Small Cell Lung Cancer (NSCLC)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3101 (Experimental): TQ-B3101 300 mg given orally in fasting conditions, twice daily in 28-day cycle.
  Interventions: Drug: TQ-B3101

INTERVENTIONS:
Drug: TQ-B3101 — TQ-B3101 300 mg given orally in fasting conditions, twice daily in 28-day cycle.

SUMMARY:
To assess efficacy and safety of oral TQ-B3101 administered to patients with Advanced Non-Small Cell Lung Cancer (NSCLC) that confirmed ROS1 positive gene mutation.

ELIGIBILITY:
Inclusion Criteria:

1.18 years and older. 2.Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1；Life expectancy ≥ 3 months.

3.Understood and Signed an informed consent form. 4.Histologically or cytologically confirmed locally advanced or metastatic NSCLC .

5.Subjects in the screening period should provide a written report of ROS1 positive, or tumor histological specimens obtained at the time of diagnosis/post before enrollment are sent to the central laboratory to confirm ROS1 positive.

6. Had received no more than two chemotherapy regimens. 7.At least 1 measurable tumor lesion other than brain lesions within 28 days before first dose based on RECIST 1.1.

8.The main organs function are normally, the following criteria are met:

1. routine blood tests（no blood transfusion and blood products within 14 days）：hemoglobin（Hb）≥90g/L；absolute neutrophil count（ANC）≥1.5×109/L； platelets（PLT）≥100×109/L.
2. Blood biochemical examination: alanine transaminase（ALT）and aspartate aminotransferase（AST）≤2.5×upper limit of normal (ULN)（when the liver is invaded, ALT, and AST ≤5× upper limit of normal (ULN) ）； total bilirubin (TBIL)≤1.5×upper limit of normal (ULN)；Serum creatinine ≤ 1.5 × upper limit of normal (ULN); or creatinine clearance calculated ≥ 50ml / min (calculated according to Cockcroft-Gault formula);
3. left ventricular ejection fraction (LVEF) measured by the Cardiac echocardiography ≥ 50%.

   9.Women must meet one of the following conditions:has undergone surgical sterilization;have been menopausal at least 1 year;have fertility, the following conditions must be met;Serum pregnancy test results were negative; throughout the study period to 6 months after the last dose, agreed to adopt an approved method of contraception (for example: oral contraception, injection contraception or implanted, barrier-effect Contraceptive methods, spermicides and condoms, or intrauterine devices).Men must meet one of the following conditions:has surgical sterilization;an approved method of contraception must be used throughout the study period and 6 months after the last dose.

   Exclusion Criteria:
   1. Has any known endothelial growth factor receptor (EGFR) positive mutation.
   2. Prior therapy with crizotinib, anti-programmed cell death (PD)-1, anti-PD-L1 or any other ROS1 inhibitor.
   3. Has multiple factors affecting oral medication, such as inability to swallow, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.
   4. Has diagnosed and/or treated additional malignancy within 5 years prior to randomization with the exception of cured carcinoma in situ of the cervix、 non-melanoma skin cancers and superficial bladder tumors.
   5. Has a history of hypertensive crisis, hypertensive encephalopathy; or uncontrolled hypertension.
   6. Has clinically significant, uncontrolled cardio-cerebral vascular disease.
   7. Has major surgery and anti-tumor treatment before two weeks of treatment and participated in other drug clinical trials within four weeks.
   8. Has known central nervous system metastasis and/or spinal cord compression, cancerous meningitis, and pia mater disease.
   9. Has in screening period confirmed HCV positive, HIV positive, active syphilis positive, or HBsAg positive, HBV DNA titers >500 copies/ml and stable time <14 days after symptomatic treatment,or has a history of stem cells and organ transplantation.
   10. Has history of psychotropic substance abuse that unable to abstain from or mental disorder.
   11. According to the judgement of the researchers, there are other factors that may lead to the termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to approximately 20 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR).

SECONDARY OUTCOMES:
Duration of Response (DOR) | up to approximately 20 months
  DOR was defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression or to death due to any cause, whichever occurred first.
Disease control rate (DCR) | up to approximately 20 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Progression-free survival (PFS) | up to approximately 20 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | up to approximately 24 months
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Anhui chest hospital, Hefei, Anhui
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Tumor hospital, Chinese academy of medical sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Tumor Hospital, Fuzhou, Fujian
  - Affiliated tumor hospital of sun yat-sen university, Guangzhou, Guangdong
  - The first affiliated hospital of guangdong pharmaceutical university, Guangzhou, Guangdong
  - The first affiliated hospital of guangzhou medical college, Guangzhou, Guangdong
  - Affiliated tumor hospital of Harbin medical university, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Hunan provincial tumor hospital, Changsha, Hunan
  - Xiangya Hospital of Centre-south University, Changsha, Hunan
  - Second hospital of jilin university, Changchun, Jilin
  - The second affiliated hospital of dalian medical university, Dalian, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Linyi tumor hospital, Linyi, Shandong
  - Qingdao University Medical College Hospital, Qingdao, Shandong
  - Shanghai Jiaotong University Affiliated Chest Hospital, Shanghai, Shanghai Municipality
  - The first affiliated hospital of xi 'an jiaotong university, Xi’an, Shanxi
  - Tianjin tumor hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital School of Medical,Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Lu S, Pan H, Wu L, Yao Y, He J, Wang Y, Wang X, Fang Y, Zhou Z, Wang X, Cai X, Yu Y, Ma Z, Min X, Yang Z, Cao L, Yang H, Shu Y, Zhuang W, Cang S, Fang J, Li K, Yu Z, Cui J, Zhang Y, Li M, Wen X, Zhang J, Li W, Shi J, Xu X, Zhong D, Wang T, Zhu J. Efficacy, safety and pharmacokinetics of Unecritinib (TQ-B3101) for patients with ROS1 positive advanced non-small cell lung cancer: a Phase I/II Trial. Signal Transduct Target Ther. 2023 Jun 30;8(1):249. doi: 10.1038/s41392-023-01454-z. PMID 37385995